CLINICAL TRIAL: NCT01651936
Title: A Phase IIa, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter, Worldwide, Proof-of-Concept Clinical Trial to Evaluate the Safety, Tolerability, and Efficacy of MK-8457 in Subjects With Active Rheumatoid Arthritis and an Inadequate Response or Intolerance to Anti-TNF-α Therapy
Brief Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Trial to Evaluate the Safety, Tolerability, and Efficacy of MK-8457 in Participants With Rheumatoid Arthritis (MK-8457-010)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8457-010; 2012-002181-12 (EudraCT Number)
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Base Study: MK-8457 (Experimental): Participants received MK-8457 100 mg dosed twice daily (BID) orally with MTX at the stable dose received upon study enrollment. The Base Study lasted up to 24 weeks.
  Interventions: Drug: MK-8457 100 mg; Drug: Methotrexate
- Base Study: Placebo (Placebo Comparator): Participants received placebo BID orally with MTX at the stable dose received upon study enrollment. The Base Study lasted up to 24 weeks.
  Interventions: Drug: Methotrexate; Drug: Dose-match placebo
- Safety Extension: MK-8457 (Experimental): Participants received MK-8457 100 mg dosed twice daily (BID) orally with MTX at the stable dose received upon study enrollment. The Safety Extension was to last up to 76 weeks.
  Interventions: Drug: MK-8457 100 mg; Drug: Methotrexate

INTERVENTIONS:
Drug: MK-8457 100 mg — MK-8457 100 mg dosed orally BID
  Arms: Base Study: MK-8457; Safety Extension: MK-8457
Drug: Methotrexate — MTX dosed at the stable dose received upon study entry
  Other Names: Rheumatrex; Trexall
Drug: Dose-match placebo — Dose-matched placebo dosed orally BID
  Arms: Base Study: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of MK-8457 + Methotrexate (MTX) in participants with active rheumatoid arthritis (RA) and an inadequate response or intolerance to anti-tumor necrosis factor α (anti-TNF-α) therapy. The primary hypothesis of this study is that among participants with active RA, MK-8457 100 mg twice daily (BID) + MTX will be superior to placebo + MTX as measured by the change in Disease Activity Score 28 C-Reactive Protein (DAS28-CRP) after 12 weeks of treatment.

DETAILED DESCRIPTION:
In the Base Study, participants were to receive blinded MK-8457 100 mg + MTX or matched placebo + MTX for up to 24 weeks. At Week 12 and 18, efficacy evaluation was conducted to assess eligibility for early escape, defined as <20% improvement in tender and swollen joint counts. Participants who completed the Base Study and those eligible for early escape could enroll in the 76-week Safety Extension in which participants were to receive open-label MK-8457 100 mg BID + MTX.

All participants must have been treated with MTX for at least 3 months prior to Screening and have been receiving a stable dose of MTX for at least 4 weeks prior to Screening. In addition, each participant must have either failed treatment with 1 or 2 anti-TNF-α therapies or was intolerant to anti-TNF-α therapy prior to Screening. For participants who failed therapy, the treatment with anti-TNF-α therapies must have been for at least 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis for at least 6 months prior to screening
* Active rheumatoid arthritis as defined by the presence of >= 6 swollen joints (of 66 count) and >= 6 tender joints (of 68 joint count)
* C-reactive protein blood level >0.9 mg/dL or an elevated erythrocyte sedimentation rate (ESR) >28 mm/hr and evidence of synovitis on imaging
* American College of Rheumatology Functional Class I, II, or III
* Received methotrexate for a minimum of 3 months prior to screening with a regionally appropriate stable weekly dose for at least 4 weeks prior to screening. The dose of methotrexate must remain stable through Week 24 of the study.
* Failed treatment with 1 or 2 anti-tumor necrosis factor alpha (anti-TNF-α) therapies or was intolerant to anti-TNF-α therapy prior to screening
* If using non-steroidal anti-inflammatory drugs or other analgesics, participant must be on a stable dose
* No history of either untreated latent or active tuberculosis (TB) prior to baseline
* Participants of reproductive potential must agree to remain abstinent or use 2 acceptable methods of birth control

Exclusion Criteria:

* Presence of inflammatory disease other than rheumatoid arthritis, including but not limited to psoriatic arthritis, ankylosing spondylitis, systemic lupus erythematosus, or Lyme disease
* Hospitalization due to an acute cardiovascular event, cardiovascular illness, or cardiovascular surgery within 6 months of screening
* Participant has a transplanted organ, excluding corneal transplant, performed > 3 months prior to the first dose of trial medication
* History of, or current ongoing ,chronic or recurrent infectious disease
* Positive hepatitis B surface antigen or hepatitis C test result
* Human immunodeficiency virus (HIV) positive
* User of recreational or illicit drugs or has had a history (within the previous 2 years) of drug or alcohol abuse or dependence
* Prior exposure to fostamatinib or other spleen tyrosine kinase inhibitors
* Prior exposure to 3 or more anti-TNF therapeutic agents
* Has been treated for RA with a marketed biologic agent (other than anti-TNF therapeutic agents) and failed the agent due to lack of efficacy
* Currently participating in another interventional clinical trial or has participated in an interventional clinical trial within 4 weeks prior to screening
* Severe opportunistic infection within the 6 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-08-29 (Actual); Primary Completion 2013-10-08 (Actual); Study Completion 2013-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 53 clinical centers in the United States, Australia, Columbia, Denmark, France, Greece, Hungary, Italy, New Zealand, Poland, South Africa, Spain, and in the United Kingdom. A total of 120 participants were screened and 56 were enrolled.
Groups:
- Base Study: MK-8457: MK-8457 100 mg BID + MTX for up to 24 weeks in the Base Study
- Base Study: Placebo: Placebo BID + MTX for up to 24 weeks in the Base Study
- Extension Study: MK-8457: MK-8457 100 mg BID + MTX for up to 76 weeks in the Extension Study. Participants who completed or had early escape from the Base Study were eligible to enroll in the Extension Study.
Period: Base Study
Arm/Group | Base Study: MK-8457 | Base Study: Placebo | Extension Study: MK-8457
Started | 30 | 26 | 0
Completed | 3 | 1 | 0
Not Completed | 27 | 25 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Early Escape | 2 | 8 | 0
Not completed — Study terminated by sponsor | 21 | 16 | 0
Period: Extension Study
Arm/Group | Base Study: MK-8457 | Base Study: Placebo | Extension Study: MK-8457
Started | 0 | 0 | 14 (Includes completers and early escapees from the Base Study)
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 14
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 13

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Base Study: MK-8457 | Base Study: Placebo | Total
Number analyzed (Participants) | 30 | 26 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.8 (12.7) | 59.3 (10.8) | 58.5 (11.8)
Age, Customized [Number; unit: Participants]
  <65 years | 21 | 20 | 41
  ≥65 years | 9 | 6 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score (DAS28) as Measured by C-Reactive Protein (CRP) at Week 12
Description: The DAS28-CRP is a continuous parameter based upon a statistically-derived index combining tender joints (28 joints; 0=absent, 1=present; TEN28), swollen joints (28 joints; 0=absent, 1=present; SW28), CRP (an inflammatory marker, decrease indicates improvement), and Patient's Global Assessment of Disease Activity Visual Analog Scale (VAS) (0=doing very well to 100=doing very poor; GH). It is defined as follows: DAS28-CRP = 0.56 × SQRT(TEN28) + 0.28 × SQRT(SW28) + 0.36 × ln (CRP+1) + 0.014 × GH + 0.96. The DAS28-CRP is a scale ranging from 0 to 10 with higher values indicating greater RA disease activity. This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 12
Population: Randomized participants in the Base Study who received at least one dose of study drug and had both Baseline and Week 12 DAS28-CRP measurements
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Base Study: MK-8457 | Base Study: Placebo
Number analyzed (Participants) | 13 | 18
Units on a scale | -1.83 [-2.58 to -1.09] | -1.31 [-2.01 to -0.62]
Statistical Analysis 1: Comparison: Base Study: MK-8457 vs Base Study: Placebo; Test type: Superiority or Other; p = 0.308, Constrained Longitudinal Data Analysis; Difference in least squares means = -0.52, 95% CI 2-sided [-1.54 to 0.50]

2. Secondary Outcome: Percentage of Participants Achieving an American College of Rheumatology (ACR) 20 Response at Week 12
Description: ACR responses are numerical measurements of improvement in multiple disease assessment criteria. An ACR20 response is defined as a ≥20% improvement in 1) swollen joint count (66 joints) and tender joint count (68 joints) (0 = Absent; 1 = Present) and 2) ≥20% improvement in 3 of the following 5 assessments: a) a participant's overall assessment of pain on a visual analog scale (VAS, no pain =0 to extreme pain =100); b) Patient's Global Assessment of Disease Activity VAS (doing very well =0 to doing very poor =100); c) Investigator's Global Assessment of Disease Activity VAS (doing very well =0 to doing very poor =100 ; d) participant's assessment of function across 8 functional areas as measured by Health Assessment Questionnaire (HAQ), total scores ranging from no difficulty =0 to inability to perform tasks =24; and e) serum C-Reactive Protein (decrease indicates improvement). This outcome measure applied to Base Study participants only.
Time Frame: Week 12
Population: Randomized participants in the Base Study who received at least one dose of study drug and had at least one post-baseline ACR20 measurement (last observation carried forward)
Measure: Number; unit: Percentage of participants
Arm/Group | Base Study: MK-8457 | Base Study: Placebo
Number analyzed (Participants) | 30 | 26
Percentage of participants | 26.67 | 26.92
Statistical Analysis 1: Comparison: Base Study: MK-8457 vs Base Study: Placebo; Test type: Superiority or Other; p = 0.91, Cochran-Mantel-Haenszel; Difference in percentages = -0.26, 95% CI 2-sided [-23.52 to 23.01]

3. Secondary Outcome: Percentage of Participants Achieving an ACR20 Response at Week 24
Description: as for outcome 2
Time Frame: Week 24
Population: Due to the early termination of the study, analysis for this outcome measure was not performed according to the protocol because complete data were not available.
Arm/Group | Base Study: MK-8457 | Base Study: Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants Achieving an ACR50 Response at Week 12
Description: ACR responses are numerical measurements of improvement in multiple disease assessment criteria. An ACR50 response is defined as a ≥50% improvement in 1) swollen joint count (66 joints) and tender joint count (68 joints) (0 = Absent; 1 = Present) and 2) ≥50% improvement in 3 of the following 5 assessments: a) a participant's overall assessment of pain on a visual analog scale (VAS, no pain =0 to extreme pain =100); b) Patient's Global Assessment of Disease Activity VAS (doing very well =0 to doing very poor =100); c) Investigator's Global Assessment of Disease Activity VAS (doing very well =0 to doing very poor =100 ; d) participant's assessment of function across 8 functional areas as measured by Health Assessment Questionnaire (HAQ), total scores ranging from no difficulty =0 to inability to perform tasks =24; and e) serum C-Reactive Protein (decrease indicates improvement). This outcome measure applied to Base Study participants only.
Time Frame: Week 12
Population: Randomized participants in the Base Study who received at least one dose of study drug and had at least one post-baseline ACR50 measurement (last observation carried forward)
Measure: Number; unit: Percentage of participants
Arm/Group | Base Study: MK-8457 | Base Study: Placebo
Number analyzed (Participants) | 30 | 26
Percentage of participants | 20.00 | 11.54
Statistical Analysis 1: Comparison: Base Study: MK-8457 vs Base Study: Placebo; Test type: Superiority or Other; p = 0.468, Cochran-Mantel-Haenszel; Difference in percentages = 8.46, 95% CI 2-sided [-10.40 to 27.32]

5. Secondary Outcome: Change From Baseline in DAS28-CRP at Week 24
Description: The DAS28-CRP is a continuous parameter based upon a statistically-derived index combining tender joints (28 joints; 0=absent, 1=present; TEN28), swollen joints (28 joints; 0=absent, 1=present; SW28), CRP (decrease indicates improvement), and Patient's Global Assessment of Disease Activity Visual Analog Scale (VAS) (0=doing very well to 100=doing very poor; GH, ). It is defined as follows: DAS28-CRP = 0.56 × SQRT(TEN28) + 0.28 × SQRT(SW28) + 0.36 × ln (CRP+1) + 0.014 × GH + 0.96. The DAS28-CRP is a scale ranging from 0 to 10 with higher values indicating greater RA disease activity. This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 24
Population: as for outcome 3
Arm/Group | Base Study: MK-8457 | Base Study: Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire Disability (HAQ Disability Index) at Week 12
Description: The functional status of the participant was assessed using the Disability Index of the HAQ on a Likert scale. This 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area. The overall score for the Disability Index is the mean of the 8 functional area scores and also ranges from 0 to 3, with a lower score indicating less disability. A negative change from Baseline indicates improvement. This outcome measure applied to Base Study participants only.
Time Frame: Baseline and Week 12
Population: Randomized participants in the Base Study who received at least one dose of study drug and had both Baseline and Week 12 HAQ Disability Index measurement
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Base Study: MK-8457 | Base Study: Placebo
Number analyzed (Participants) | 13 | 18
Units on a scale | -0.67 [-0.95 to -0.39] | -0.26 [-0.52 to -0.01]
Statistical Analysis 1: Comparison: Base Study: MK-8457 vs Base Study: Placebo; Test type: Superiority or Other; p = 0.038, Constrained Longitudinal Data Analysis; Difference in least squares means = -0.41, 95% CI 2-sided [-0.79 to -0.02]

7. Secondary Outcome: Percentage of Participants Achieving an ACR50 Response at Week 24
Description: ACR responses are numerical measurements of improvement in multiple disease assessment criteria. An ACR50 response is defined as a ≥50% improvement in 1) swollen joint count (66 joints) and tender joint count (68 joints) (0=Absent; 1=Present) and 2) ≥50% improvement in 3 of the following 5 assessments: a) a participant's overall assessment of pain on a visual analog scale (VAS, 0=no pain to 100=extreme pain); b) Patient's Global Assessment of Disease Activity VAS (0=doing very well to 100=doing very poor); c) Investigator's Global Assessment of Disease Activity VAS (0=doing very well to 100=doing very poor; d) participant's assessment of function across 8 functional areas as measured by Health Assessment Questionnaire (HAQ), total scores ranging from 0=no difficulty to 24=inability to perform tasks; and e) CRP (decrease indicates improvement). This outcome measure applied to Base Study participants only.
Time Frame: Week 24
Population: as for outcome 3
Arm/Group | Base Study: MK-8457 | Base Study: Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in the HAQ Disability Index at Week 24
Description: as for outcome 6
Time Frame: Baseline and Week 24
Population: as for outcome 3
Arm/Group | Base Study: MK-8457 | Base Study: Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Base Study: up to 24 weeks: Extension Study: up to approximately 40 weeks
Arm/Group | Base Study: MK-8457 | Base Study: Placebo | Extension Study: MK-8457
Serious Adverse Events (participants affected / at risk) | 5/30 | 0/26 | 2/14
Other Adverse Events (participants affected / at risk) | 10/30 | 2/26 | 6/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study: MK-8457 (N=30) | Base Study: Placebo (N=26) | Extension Study: MK-8457 (N=14)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study: MK-8457 (N=30) | Base Study: Placebo (N=26) | Extension Study: MK-8457 (N=14)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early (12 September 2013) based on preliminary analysis of data. The results of this study need to be interpreted with caution given the small sample size (56 participants) resulting from early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.